CLINICAL TRIAL: NCT05392478
Title: The Effects of Body Mass İndex On İntraabdominal Pressure And Regional Cerebral Oxygen Saturation İn Lumbar Spine Surgery İn Prone Position
Brief Title: The Effects of Body Mass İndex On İntraabdominal Pressure And Regional Cerebral Oxygen Saturation İn Prone Position
Status: Completed | Type: Observational
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ozlem Sen, MD, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Other Study IDs: 2182NIRS
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Cerebral Hypoxia During and/or Resulting From A Procedure
Keywords: cerebral oxygenation, prone position, obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A total of 40 ASA (American Society of Anesthesiology) physical status I-III who underwent lumbar disc hernia repair for one or two levels were included in this prospective study. A standard anesthesia protocol was performed in all patients. Routine intraoperative monitoring consisted of electrocardiography, automatic noninvasive arterial blood pressure, pulse oximetry, capnography, and cerebral tissue oxygen saturation through NIRS.Patients' demographics such as age, gender, height, weight, BMI, smoking status and pre-existing medical conditions were recorded.The patients were allocated equally to two groups according to BMI as Group I: BMI ≥30kg/m2,Group II <30 kg/m2.

DETAILED DESCRIPTION:
Routine intraoperative monitoring consisted of electrocardiography, automatic noninvasive arterial blood pressure, pulse oximetry, capnography, and cerebral tissue oxygen saturation through NIRS.Frontal lobe oxygenation was monitored continuously and recorded every 5 minutes.Before positioning patients on the operating table, a Foley catheter was placed. IAP was measured in the following positions in all patients: 1) in the supine position after intubation 2) in the prone position before the skin incision.All patients were placed into the prone position on the silicone pads after general anesthesia.Before statistical analysis, the 40 patients were allocated equally to two groups according to the World Health Organization Guideline of BMI: Group I: BMI ≥30kg/m2, Group II <30 kg/m2

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* ASA physical status I - III patients undergoing lumbar disc hernia repair for two or less levels

Exclusion Criteria:

* Age smaller than 18 or older than 70 years,
* ASA physical status more than III,
* Patients with a history of carotid artery stenosis, prior neck surgery, cervical canal stenosis, stroke, neurological deficit, myocardial infarction, spinal cord injury and sudden vision loss

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 40 ASA physical status I - III patients undergoing lumbar disc hernia repair for two or less levels. The ethical committee approval for the study was taken from the Abdurrahman Yurtaslan Oncology Training and Research Hospital (2014-2182). The informed consent was obtained for all the patients that were included in the study
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-03-10 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Cerebral tissue oxygen saturation with NIRS .Effect os boddy mass index on cerebral tissue oxygen saturation in prone position | İntraoperatif ( During surgery)
  Effects of boddy mass index and intraabdominal pressure on cerebral tissue oxygen saturation in prone position

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Şen, Principal Investigator — Trabzon Kanuni Training and Research Hospital; Dilek Kalaycı, Study Chair — Dr.Abdurrahman Yurtaslan Oncology Training and Research Hospital; Süheyla Ünver, Study Chair — Dr.Abdurrahman Yurtaslan Oncology Training and Research Hospita; Tülay Dal, Study Chair — Dr.Abdurrahman Yurtaslan Oncology Training and Research Hospita; Kübra Kutay, Study Chair — Bağcılar Training and Research Hospital